Version 1.0 Statistical Reporting and Analysis plan, 27 Feb 2018



# STATISTICAL REPORTING AND ANALYSIS PLAN

A single dose, open label, randomized scintigraphic study to investigate the gastrointestinal behavior of 2 triple combination products (Acetaminophen, Phenylephrine and Dextromethorphan) in healthy male volunteers

Protocol Number: 208821

Phase: 1

Property of GSK Consumer Healthcare
Confidential
May not be used, divulged, published or otherwise disclosed
without the consent of GSK
Template Version Effective: 15-Jul-2017


# **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Original Analysis Plan | 27-Feb-2018 | Not applicable (N/A) |

Amendments incorporate all revisions to date.

#### Table of contents Document History......2 Abbreviation ......5 Summary of Key Protocol Information ......6 1.1 Study Design.....6 1.2 Study Objectives ......6 1.3 1.4 Planned Analyses ......8 2.1 Interim Analysis......8 2.2 3 Considerations for data analyses and Data Handling Conventions ......8 3.1 Baseline Definition ......8 3.2 Centers Pools......8 3.3 3.4 Timepoints and Visit Windows.....8 Data Analysis ......9 4.1 Populations for Analysis ......9 4.1.1 Subject Disposition......9 4.1.2 4.1.3 4.2 4.2.1 4.2.2 General Medical History ......11 Treatments (Study Treatment, Rescue Medication, other Concomitant 4.3 Therapies, Compliance)......11 4.3.1 Study Treatment Compliance and Exposure ......11 4.3.2 Analysis of Efficacy......11 4.4 4.4.1 4.4.2 Secondary Efficacy Variables ......12 4.4.3

GlaxoSmithKline Consumer Healthcare Confidential


| | 4.5 | Analys | is of Gamma Scintigraphy Imaging | 12 |
|-----|------|------------|----------------------------------------------|----|
| | 4.6 | Analys | is of Safety | 13 |
| | | 4.6.1 | Adverse Events and Serious Adverse Events | 13 |
| | | 4.6.2 | Laboratory Tests | 13 |
| | | 4.6.3 | Vital Signs | 13 |
| | | 4.6.4 | Findings on Physical Examination | |
| | | 4.6.5 | Electrocardiogram | 14 |
| | | 4.6.6 | Other Safety Variables | 14 |
| | 4.7 | Analys | is of Other Variables | |
| | | 4.7.1 | Quality of Life | 14 |
| | | 4.7.2 | Patch Adhesion Performance | 14 |
| 5 | Chan | ges to the | e Protocol Defined Statistical Analysis Plan | 14 |
| Att | | _ | of Data Displays | |
| 6 | | | emplate for Tables, Figures and Listings | |


# **Abbreviation**

| Abbreviation | Term |
|--------------|----------------------------------------------|
| AE | Adverse Event |
| AUC | Area Under the Curve |
| BMI | Body Mass Index |
| DRM | Data Review Meeting |
| CI | Confidence Interval |
| CV | Coefficient of Variation |
| ECG | Electrocardiogram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| soc | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |


The purpose of this Statistical Reporting and Analysis Plan is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 208821 (v2.0 dated 25 Jan 2018).

# 1 Summary of Key Protocol Information

This clinical study will be conducted to characterize the gastrointestinal transit of two multisymptom formulations by inclusion of a radiolabel marker: Theraflu Daytime Severe Cold and Cough powder for oral solution and Theraflu ExpressMax Daytime Severe Cold and Cough caplets.

This study will be the first study to investigate the time of onset and completion of gastric emptying as well as small intestine transit time of Theraflu Daytime Severe Cold and Cough powder for oral solution and Theraflu ExpressMax Daytime Severe Cold and Cough caplets.

# 1.1 Study Design

This will be an open label, randomized, single dose, and parallel group gamma scintigraphy. Approximately, forty-two healthy male volunteers will be screened to allow a total of 28 healthy male volunteers to be randomized (14 subjects per treatment group) in order to have 24 evaluable subjects (12 subjects per treatment group).

Subjects will be randomized to receive either a single dose of Theraflu Daytime Severe Cold and Cough powder for oral solution (Treatment A) or a single dose of Theraflu ExpressMax Daytime Severe Cold and Cough caplets (Treatment B) under fasted conditions:

Treatment A - 12 healthy male volunteers will be administered 1 sachet of Theraflu Daytime Severe Cold and Cough radiolabeled powder for oral solution (acetaminophen 650 mg + phenylephrine 10 mg + 20 mg dextromethorphan) reconstituted with 225 mL of hot water.

Treatment B-12 healthy male volunteers will take 2 radiolabeled caplets of Theraflu ExpressMax Daytime Severe Cold and Cough (2 caplets each containing acetaminophen 325 mg + phenylephrine 5 mg + 10 mg dextromethorphan) with 225 mL of room temperature noncarbonated water.

# 1.2 Study Objectives

The study objectives are as follows:

| Objectives | Endpoints |
|---|---|
| Gamma Scintigraphy Imaging | |
| Characterize time to onset and time to completion | Mean time to onset of gastric emptying in healthy |
| of gastric emptying after administration of either | male volunteers who did not vomit shortly (within 60 |
| Theraflu Daytime Severe Cold and Cough | minutes) after study drug administration, who have |
| powder for oral solution to be reconstituted with | sufficient data to determine time to onset of gastric |


| Objectives | Endpoints |
|---|---|
| 225 ml of hot water or Theraflu ExpressMax | emptying and who had no major protocol deviations. |
| Daytime Severe Cold and Cough caplets using | Mean time to complete gastric emptying in healthy |
| gamma scintigraphic analysis. | male volunteers who did not vomit shortly (within 60 |
| | minutes) after study drug administration, who have |
| | sufficient data to determine time to completion of |
| | gastric emptying and who had no major protocol deviations. |
| | Further characterize gastrointestinal emptying (GE) by calculating additional parameters such as but not limited to: a) GE25%, GE50%, GE90% values, b) the amount remaining in the stomach at 15, 30, 45, 60, 75, 90, 105, 120, 180, 240 min; c) sectional areas under the gastric emptying curve (AUC) and total AUC; and d) gastric emptying t <sub>1/2</sub> values. e) Small intestinal transit times which are calculated by determining the arrival time of the radioactive marker at the cecum / colon region and subtracting the gastric emptying value. |
| C - C | |
| Safety | |
| To evaluate safety of Theraflu Daytime Severe | A safety assessment consists of monitoring and |
| Cold and Cough powder for oral solution and | recording adverse events (AEs) and laboratory test. |
| Theraflu ExpressMax Daytime Severe Cold and | |
| Cough caplets | |

#### 1.3 Treatments

The healthy male individuals will be randomized to take either of the following two treatments:

**Treatment A:** 1 sachet of Theraflu Daytime Severe Cold and Cough powder (Berry flavor) - (acetaminophen 650mg + Dextromethorphan 20mg + Phenylephrine 10mg).

**Treatment B:** 2 caplets of Theraflu ExpressMax Daytime Severe Cold and Cough (each caplet contains: acetaminophen 325 mg + Dextromethorphan 10mg + Phenylephrine 5mg).

Both products will be commercially sourced from local market.

#### 1.4 Sample Size Calculation

Since this study does not have any statistical power, formal sample size calculation has not been performed. It is planned to screen approximately 42 subjects to allow a total of 28 subjects to be randomized to have at least 24 subjects evaluable (12 subject per treatment group). This is a sufficient number to provide descriptive statistics.


# 2 Planned Analyses

#### 2.1 Interim Analysis

No interim analysis is planned.

# 2.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- All subjects have completed the study as defined in the protocol.
- All required database cleaning activities have been completed and database has been locked.

# 3 Considerations for data analyses and Data Handling Conventions

#### 3.1 Baseline Definition

A baseline definition is not required for this study as no baseline measurements are performed or required for the summaries and analysis.

#### 3.2 Subgroups/Stratifications

No subgroups or stratifications factors are defined in this study.

#### 3.3 Centers Pools

Since this is single center study, pooling of centres is not applicable.

# 3.4 Timepoints and Visit Windows

The study will consist of screening visit (Visit 1), followed by a treatment visit (Visit 2). Visit 2 includes two days: Day -1 and Day 1. The screening visit will assess subject eligibility and consist of relevant medical examinations.

On Visit 2 (Day -1) of the study, subjects will be admitted to the unit at approximately 7 pm on the evening before study drug administration to ensure compliance with fasting conditions and will receive a standardized meal. Subjects are required to fast (nothing to eat or drink except room temperature non-carbonated water) from 10 hours prior until 4 hours after study drug administration. Water is permitted until 1 hour prior to investigational product administration, and no additional fluids until the lunch meal is served at approximately 4 hours post dose.


Subjects will be given a standard lunch at 4 hours post-dose and a standard dinner at 10 hours post-dose on Day 1. Subjects will be discharged from the unit after the last scintigraphic imaging is performed; blood sample for laboratory test is taken as well as a brief physical examination.

The timepoints and visits for this study are defined in the section "Schedule of Activities" of the protocol. Any deviation from the study schedule will be reviewed on case-by-case basis to determine whether the data should be excluded from any analysis. A time window non-compliance listing will be produced for the Data Review Meeting (DRM).

# 4 Data Analysis

Data analysis will be performed by Syneos Health. The statistical analysis software used will be SAS version 9.4 (Studio) or higher.

Prior to database closure a DRM will be conducted in which various aspects of the study will be discussed and agreed.

Unless otherwise described below, all listings will be produced for all randomized subjects.

# 4.1 Populations for Analysis

### 4.1.1 Subject Disposition

Screen failures will be defined as subjects who do not satisfy either of the inclusion or exclusion criteria and are not subsequently randomized. A summary table for number of subjects screened, number of screen failure subjects with reasons why not randomized (Table 14.1.1) will be presented. The percentage will be based on total number of screened subjects.

Subject disposition will also be summarized as the number and percentage of subjects in each of the defined analysis population, who complete the study, who discontinue the study and reason for discontinuation (Table 14.1.1). The summary table will be presented by each treatment group and for all combined treatment group (Overall). The percentage will be based on total number of subjects randomized in each treatment and overall.

Subject disposition including the critical demographic data (age and sex), screening date, date and time of treatment administration, date of completion or withdrawal, subject status (completer, Yes/No) and the specific reason for discontinuation, will be listed in Listing 16.2.1.1 by treatment groups for randomized subjects and non-randomized subjects (Listing 16.2.1.2) separately.

#### 4.1.2 Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study. Data will be reviewed at DRM prior to closure of the database to ensure all important deviations are captured and categorized.

GlaxoSmithKline Consumer Healthcare Confidential


Major deviations of the protocol procedures identified as liable to influence the outcome of the study may include, but will not be necessarily limited to the following:

- Inclusion/Exclusion criteria
- Treatment administration error
- Use of prohibited medications before and during the study which is deemed to affect the assessment of efficacy
- Deviations likely to affect study outcomes
- Vomiting shortly (within 60 minutes) after study drug administration

The number and percentage of subjects with any major protocol deviations and with each type of major protocol deviations will be presented by treatment (Table 14.1.2) and listed in Listing 16.2.2.1. Any minor protocol deviations will be listed similarly (Listing 16.2.2.2).

#### 4.1.3 Analysis Populations

In this study following analysis populations are defined:

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety Population | All subjects who receive a radiolabeled treatment A or | Safety Analysis |
| | B irrespective of whether the subject is included in the | |
| | scintigraphy analysis. | |
| Scintigraphy | All subjects who receive the radiolabeled treatment A | Scintigraphy Analysis |
| Analysis | and B and who did not vomit shortly (within 60 | |
| Population | minutes) after the study drug administration, who have | |
| | sufficient data to determine time to onset and | |
| | completion of gastric emptying and who had no major | |
| | protocol deviations. | |

#### NOTES:

• Please refer to Attachment 1: List of Data Displays which details the population to be used for each displays being generated.

Subjects excluded from any of the analysis populations will be listed in Listing 16.2.3.1, with the reason for exclusion.

# 4.2 Subject Demographics and Other Baseline Characteristics

Demographic and baseline summarizes will be produced for all subjects in safety population.

#### 4.2.1 Demographic Characteristics

Descriptive statistics [number of subjects (n), mean, standard deviation (SD), median, minimum and maximum values] for continuous variables and frequency count (n) and percentages (%) for all categorical variables will be presented.


The demographic characteristic includes age (in years) and height (in cm). This data will be summarized descriptively for all subjects in safety population (Table 14.1.3) by treatment group and overall and will be listed (Listing 16.2.4.1) for all randomized subjects.

#### 4.2.2 General Medical History

Medical history will be listed in Listing 16.2.4.2, with start date and end date or ongoing at the start of study drug.

# 4.3 Treatments (Study Treatment, Rescue Medication, other Concomitant Therapies, Compliance)

#### 4.3.1 Study Treatment Compliance and Exposure

Study treatment will be administered under the supervision of investigator site personnel and hence the summary and listing will not be required.

#### 4.3.2 Prior and Concomitant Medication

Prior or concomitant medication taken by or administered to a subject will be recorded in the case report form. The prior and concomitant medications will be coded using an internal validated medication dictionary, GSKDrug.

Prior medication will be listed by subject, with drug name, GSK drug synonym, dose, reason for medication, route, dose frequency start date, study day relative to study treatment administration and end date (Listing 16.2.5.1). Prior medications are defined as medications that are stopped before study treatment administration. If the start or stop date is unknown or incomplete and medication cannot be considered as stopped prior to first administration of study treatment then the medication will be considered as concomitant medication.

Concomitant medications will be listed similarly (Listing 16.2.5.2) with either ongoing or end date displayed. Concomitant medications are defined as the medications ongoing or started after the study treatment administration.

Unknown dates will not be imputed, however if the start or stop date is unknown, then it will be assumed to a concomitant medication, unless the partial start date or stop date indicates differently.

# 4.4 Analysis of Efficacy

No applicable as there are no efficacy assessments.

#### 4.4.1 Primary Efficacy Endpoint

No applicable.

GlaxoSmithKline Consumer Healthcare Confidential


#### 4.4.1.1 Primary Efficacy Endpoint Definition

No applicable.

## 4.4.1.2 Statistical Hypothesis, Model, and Method of Analysis

No applicable.

### 4.4.2 Secondary Efficacy Variables

In this study secondary efficacy variables are not defined.

# 4.4.3 Handling of Missing Values/Censoring/Discontinuations

Subjects who drop out will not be replaced and missing data will not be imputed. Dropouts will be included in analyses up to the point of discontinuation.

# 4.5 Analysis of Gamma Scintigraphy Imaging

The scintigraphy variables are:

- Time to onset of gastric emptying for treatment A and B.
- Time to completion of gastric emptying for treatment A and B.
- GE25%, GE50%, GE90% values for each treatment A and B,
- The amount remaining in the stomach at 15, 30, 45, 60, 75, 90, 105, 120, 180, 240 min for each Treatment A and B
- Sectional areas under the gastric emptying curve and total AUC; and gastric emptying  $t_{1/2}$  values.
- Small intestinal transit times for each treatment A and B.

The scintigraphic images measure the gastric emptying time to onset and completion as for treatment A and B.

The small intestinal transit times which are calculated by determining the arrival time of the radioactive marker at the cecum / colon region and subtracting the gastric emptying value.

The scintigraphy variables of scintigraphic analysis will be summarized (Table 14.2.1 – 14.2.6) by treatment group using descriptive statistics [number of subjects (n), mean, minimum, median, maximum and standard deviation, coefficient of variation (CV) and 95% confidence interval (CI) for the Means] for all subjects in scintigraphy analysis population.

Listing will be provided for the variables time to onset of gastric emptying and time to completion of gastric emptying (Listing16.2.6.1) for all subjects in scintigraphy analysis population.


The mean ( $\pm$ SD) plot across time will be presented by treatment for amount remaining in the stomach (Figure 14.2.3) and sectional areas under the gastric emptying curve (Figure 14.2.4).

There are no formal hypotheses being tested in this study.

# 4.6 Analysis of Safety

Safety variables will be summarized on all subjects in safety population

#### 4.6.1 Adverse Events and Serious Adverse Events

AEs recorded during the study will be mapped to a system organ class (SOC) and preferred term (PT) using the current medical dictionary for regulatory activities (MedDRA).

Prior to database lock all AEs will be reviewed by the Clinical Research Director (or designee).

Treatment emergent adverse events (TEAEs) are defined as AEs that start on or after study treatment administration. All AEs will be summarized by SOC and PT treatment group and overall

The following summary tables and listings will be presented by treatment group:

- Table of TEAEs by SOC and PT (Table 14.3.1.1.1)
- Table of TEAEs related to study treatment by SOC and PT (Table 14.3.1.1.2)
- Table of TEAEs by severity, SOC and PT (Table 14.3.1.2)
- Listing of all AEs (including all subjects: Listing 16.2.7.1.1 for all randomized subjects; Listing 16.2.7.1.2 for non-randomized subjects)

#### 4.6.2 Laboratory Tests

The laboratory data [Hematology, Serum Chemistry, Urinalysis, Virology (HIV antibodies, HBsAg, anti-HBc (Total), anti-HCV)] will be collected at Visit 1 and Visit 2 (Day 1) after final scintigraphic image is taken prior to dinner.

Laboratory parameters for which reference ranges will be available will then be categorized with respect to reference ranges as: High, Low, Normal and Missing.

The laboratory test results will be listed in Listings 16.2.8.1 - 16.2.8.6 and laboratory normal ranges will be listed Listing 16.2.8.7.

#### 4.6.3 Vital Signs

The vital signs data will be collected at Visit 1 and Visit 2 (Day -1 and 1). The vital signs data of systolic and diastolic blood pressure, respiratory rate, pulse rate and oral temperature


recorded at Visit 1 and Visit 2 (Day -1); whereas at Visit 2 (Day 1) blood pressure and pulse rate will be collected.

Vital signs at each assessment will be listed (Listing 16.2.9.1).

#### 4.6.4 Findings on Physical Examination

A full physical examination will include head, ears, eyes, nose, mouth, skin, and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, cardiovascular and neurological systems. The full physical examination will be performed on Visit 1 and Visit 2 (Day -1).

The brief physical examination will be focused on general appearance, the respiratory and cardiovascular systems, as well as towards subject reported symptoms. The brief physical examination will be performed on Visit 2 (Day 1).

The findings on the physical examination will be listed (Listing 16.2.9.2).

#### 4.6.5 Electrocardiogram

A standard 12 lead Electrocardiogram (ECG) will be performed at Visit 1. ECG data will be listed in Listing 16.2.9.3.

# 4.6.6 Other Safety Variables

Breath alcohol test, body weight (kg) and body mass index [BMI] (kg/m²) will be measured at Visit 1 and Visit 2 (Day -1). Body weight and BMI will be listed in Listing 16.2.9.4 and breath alcohol test in Listing 16.2.8.1.2.

### 4.7 Analysis of Other Variables

Not applicable.

#### 4.7.1 Quality of Life

Not applicable.

#### 4.7.2 Patch Adhesion Performance

Not applicable.

# 5 Changes to the Protocol Defined Statistical Analysis Plan

The changes from the originally planned statistical analysis specified in the protocol are outlined in .

#### Table 1 Changes to Protocol Defined Analysis Population

Protocol Reporting and Analysis Plan


| Protocol | Reporting and Analysis Plan | |
|---|---|---|
| Statistical Analysis Section | Statistical Analysis Plan | Rationale of Change |
| • 10.2.4 Definition of Analysis Population | • 4.1.3 Analysis Population | Added clarity to the definition and consistency across the population |
| | Safety Population | definitions. |
| Safety Population | All subjects who receive a | |
| The Safety population will include | radiolabeled treatment A or B | |
| all subjects who receive a | irrespective of whether the subject | |
| radiolabeled hot drink | is included in the scintigraphy | |
| independently if they are included | analysis. | |
| or not in the scintigraphy analysis. | | |


# **Attachment 1: List of Data Displays**




# 6 Appendix 1: Template for Tables, Figures and Listings

This is a guideline which will give the guidance of product labels that will be used for the table header and in the figures, listings and in the footnotes.

The product labels for the column headings will be as follow:

- Theraflu Powder
- Theraflu Caplets

The below footnotes will be displayed on each output

- Theraflu Powder: Theraflu Daytime Severe Cold and Cough powder for oral solution
- Theraflu Caplets: Theraflu ExpressMax Daytime Severe Cold and Cough caplets


Protocol 208821 Program Run Date: DDMMMYYYY

Table 14.1.1 Subject Disposition All Screened Subjects

Study Population: Screened Subjects (N = xx)

| | Theraflu Powder | Theraflu Caplets | Overall |
|---|---|---|---|
| | N (%) | N (%) | N (%) |
| Total subjects screened | | | xxx |
| Total Subjects Selectica | | | AAA |
| Subjects not randomized* | | | xxx (xx.x) |
| Did not meet study criteria | | | xxx (xx.x) |
| Adverse events | | | xxx (xx.x) |
| Lost to follow-up | | | xxx (xx.x) |
| Protocol violations | | | xxx (xx.x) |
| Withdrawal of consent | | | xxx (xx.x) |
| Others | | | xxx (xx.x) |
| ubjects randomized** | xxx | XXX | xxx |
| Completed study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not completed study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not meet study criteria | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Adverse events | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Safety population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Scintigraphy analysis population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

<sup>\*</sup> Percentages are based on number of screened subjects.

Program file name: xxxxxx

Programming note: List all the reasons of discontinuation mentioned eCRF.

Page x of y Source: Filename

<sup>\*\*</sup> Percentages are based on number of randomized subjects in each treatment group.


Protocol 208821 Program Run Date: DDMMMYYYY

# Table 14.1.2 Incidence of Major Protocol Deviations All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

| | Theraflu Powder (N = xxx) n (%) | Theraflu Caplets<br>(N = xxx)<br>n (%) | Overall<br>(N = xxx)<br>n (%) |
|---|---|---|---|
| Subjects with at least one major protocol deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Protocol deviations not leading to exclusion from scintigraphy analysis population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Deviation reason 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Major protocol deviations leading to exclusion from scintigraphy analysis population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Deviation reason 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Deviation reason 2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Percentages are based on number of randomized subjects in each treatment group.

Page x of y
Program: xxxxxx.sas
Source: Filename

Programming Note: This listing is based on some of the details in the population definition document.


Protocol 208821 Program Run Date: DDMMMYYYY

# Table 14.1.3 Demographics and Baseline Characteristics Safety Population

Study Population: Safety Population (N = xx)

| Theraflu Caplets | Overall |
|------------------|-----------|
| (N = xxx) | (N = xxx) |
| n (%) | n (%) |
| xx (xx.x) | xx (xx.x) |
| XX | XX |
| XX.X | XX.X |
| xx.xx | xx.xx |
| XX.X | XX.X |
| XX | XX |
| xx | xx |
| XX | xx |
| xxx.x | xxx.x |
| XXX.XX | XXX.XX |
| xxx.x | xxx.x |
| xxx | xxx |
| XXX | xxx |
| | xxx |

Percentages are based on number of subjects in safety population in each treatment group.

Page x of y
Program: xxxxxx.sas
Source: Filename


Protocol 208821 Program Run Date: DDMMMYYYY

Table 14.2.1

Summary of Time to Onset and Completion of Gastric Emptying

Scintigraphy Analysis Population

Study Population: Scintigraphy Analysis Population (N = xx)

| Damanahan (IInih) | Chariaria. | Theraflu Powder | Theraflu Caplets |
|---|---|---|---|
| Parameter (Unit) | Statistics | (N = xxx) | (N = xxx) |
| Gastric emptying onset time (min) | | | |
| Jastiic emptying onset time (min) | n<br>Migging | XXX | XXX |
| | Missing | XXX | XXX |
| | Mean | XXX.X | XXX.X |
| | SD | XXX.XX | XXX.XX |
| | CV | XXX | XXX |
| | Median | XXX.X | XXX.X |
| | Minimum | XXX | XXX |
| | Maximum | XXX | XXX |
| | 95% CI of Mean | xx.xx, xx.xx | xx.xx, xx.xx |
| Gastric emptying completion time (min) | n | xxx | xxx |
| | Missing | XXX | XXX |
| | Mean | XXX.X | XXX.X |
| | SD | XXX.XX | XXX.XX |
| | CV | XXX | xxx |
| | Median | XXX.X | xxx.x |
| | Minimum | xxx | xxx |
| | Maximum | XXX | XXX |
| | 95% CI of Mean | xx.xx, xx.xx | xx.xx, xx.xx |

Page x of y
Program: xxxxxx.sas
Source: Filename


Protocol 208821 Program Run Date: DDMMMYYYY

#### Table 14.2.2 Summary of Gastric Emptying 25%, 50% and 90% Scintigraphy Analysis Population

Study Population: Scintigraphy Analysis Population (N = xx)

| Darameter (minutes) | Statistics | Theraflu Powder | Theraflu Caplets |
|---|---|---|---|
| Parameter (minutes) | Statistics | (N = xxx) | (N = xxx) |
| Control of amounts of the Control of | _ | | |
| Gastric emptying 25% | n<br>Minaina | XXX | XXX |
| | Missing | XXX | XXX |
| | Mean | XXX.X | XXX.X |
| | SD | XXX.XX | XXX.XX |
| | CV | XXX | XXX |
| | Median | XXX.X | XXX.X |
| | Minimum | XXX | XXX |
| | Maximum | XXX | XXX |
| | 95% CI of Mean | xx.xx, xx.xx | xx.xx, xx.xx |
| Gastric emptying 50% | n | xxx | xxx |
| | Missing | XXX | XXX |
| | Mean | xxx.x | xxx.x |
| | SD | xxx.xx | xxx.xx |
| | CV | XXX | XXX |
| Gastric emptying 90% | n | xxx | xxx |
| | Missing | XXX | xxx |
| | Mean | XXX.X | xxx.x |
| | SD | XXX.XX | XXX.XX |
| | CV | XXX | XXX |

Page x of y Source: Filename

Programm: xxxxxx.sas

Programming Note: This table will continue for all other statistics as mentioned in the text.


:Program: xxxxx.sas

Protocol 208821 Program Run Date: DDMMMYYYY

Table 14.2.3

Summary of Amount Remaining in the Stomach Over Time
Scintigraphy Analysis Population

Study Population: Scintigraphy Analysis Population (N = xx)

| Parameter (Unit) | Time point | Statistics | Theraflu Powder | Theraflu Caplets $(N = xxx)$ |
|---|---|---|---|---|
| | | | (N = xxx) | (N - XXX) |
| Amount remaining in the stomach (%) | 15 min | n | xxx | XXX |
| | | Missing | XXX | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.XX | xxx.xx |
| | | CV | xxx | xxx |
| | | Median | xxx.x | xxx.x |
| | | Minimum | xxx | xxx |
| | | Maximum | xxx | xxx |
| | | 95% CI of Mean | xx.xx, xx.xx | XX.XX, XX.XX |
| | 30 min | n | xxx | xxx |
| | | Missing | xxx | XXX |
| | | Mean | XXX.X | xxx.x |
| | | SD | XXX.XX | xxx.xx |
| | 45 min | n | xxx | xxx |
| | | Missing | xxx | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.XX | XXX.XX |

Page x of y Source: Filename

Programming Note: This table will continue for all other time point and statistics as mentioned in the text.


Protocol 208821 Program Run Date: DDMMMYYYY

 ${\tt Table~14.2.4}$  Summary of Sectional Areas under the Gastric Emptying Curve Over Time Scintigraphy Analysis Population

Study Population: Scintigraphy Analysis Population (N = xx)

| Parameter (%*min) | Time point | Statistics | Theraflu Powder $(N = xxx)$ | Theraflu Caplets (N = xxx) |
|---|---|---|---|---|
| | | | , | · |
| Area under the gastric emptying curve | 15 min | n | xxx | xxx |
| | | Missing | xxx | XXX |
| | | Mean | xxx.x | xxx.x |
| | | SD | xxx.xx | xxx.xx |
| | | CV | xxx | XXX |
| | | Median | xxx.x | xxx.x |
| | | Minimum | xxx | xxx |
| | | Maximum | xxx | xxx |
| | | 95% CI of Mean | xx.xx, xx.xx | xx.xx, xx.xx |
| | 30 min | n | xxx | xxx |
| | | Missing | xxx | xxx |
| | | Mean | XXX.X | xxx.x |
| | | SD | xxx.xx | xxx.xx |
| Total area under curve | | n | xxx | xxx |
| | | Missing | xxx | xxx |
| | | Mean | xxx.x | xxx.x |
| | | SD | xxx.xx | xxx.xx |

Page x of y :Program: xxxxx.sas Source: Filename

Programming Note: This table will continue for all other time point and statistics as mentioned in the text.


Protocol 208821 Program Run Date: DDMMMYYYY

# Table 14.2.5 Summary of Gastric Emptying Half Life Scintigraphy Analysis Population

Study Population: Scintigraphy Analysis Population (N = xx)

| Parameter (min) | Statistics | Theraflu Powder (N = xxx) | Theraflu Caplets $(N = xxx)$ |
|---|---|---|---|
| Gastric emptying half life | n | xxx | xxx |
| | Missing | XXX | XXX |
| | Mean | xxx.x | xxx.x |
| | SD | xxx.xx | xxx.xx |
| | CV | XXX | XXX |
| | Median | XXX.X | xxx.x |
| | Minimum | XXX | xxx |
| | Maximum | XXX | XXX |
| | 95% CI of Mean | xx.xx, xx.xx | xx.xx, xx.xx |

Page x of y :Program: xxxxx.sas Source: Filename


Protocol 208821 Program Run Date: DDMMMYYYY

# Table 14.2.6 Summary of Small Intestinal Transit Times Scintigraphy Analysis Population

Study Population: Scintigraphy Analysis Population (N = xx)

| Parameter (min) | Statistics | Theraflu Powder | Theraflu Caplets |
|---|---|---|---|
| . , , | | (N = xxx) | (N = xxx) |
| Small intestine transit time | n | xxx | xxx |
| | Missing | XXX | xxx |
| | Mean | XXX.X | xxx.x |
| | SD | XXX.XX | XXX.XX |
| | CV | XXX | XXX |
| | Median | XXX.X | XXX.X |
| | Minimum | XXX | XXX |
| | Maximum | XXX | XXX |
| | 95% CI of Mean | xx.xx, xx.xx | XX.XX, XX.XX |

Page x of y :Program: xxxxx.sas Source: Filename


Protocol 208821 Program Run Date: DDMMMYYYY

#### 

| System Organ Class<br>Preferred Term | Theraflu Powder $(N = xxx)$ | | Theraflu Caplets<br>(N = xxx) | | Overall (N = xxx) | |
|---|---|---|---|---|---|---|
| | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| Jumber of subjects with at least one AE | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | XX |
| Number of subjects with no AE | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| System Organ Class 1 | xx (xx.x) | XX | xx (xx.x) | xx | xx (xx.x) | XX |
| Preferred Term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| System Organ Class 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

n (%) = Number (percent) of subjects; nAE = Number of adverse events. Percentages are based on number of subjects in safety population in each treatment group.

Page x of y
Program: xxxxxx.sas

Source: Filename

Programming Note: This table will continue for SOC and PT. Similar table (Table 14.3.1.1.2) will be generated for Related TEAEs by SOC and PT


Protocol 208821 Program Run Date: DDMMMYYYY

Study Population: Safety Population (N = xxx)

| | | Theraflu | Powder | Theraflu C | aplets | Overa | 11 |
|---|---|---|---|---|---|---|---|
| System Organ Class Preferred Term | Severity | (N = xxx) | | (N = xxx) | | (N = XXX) | |
| | | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| Any System Organ Class | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| | Moderate | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Severe | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| System Organ Class 1 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| | Moderate | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Severe | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 1 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Moderate | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Severe | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 2 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Moderate | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Severe | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

n (%) = Number (percent) of subjects; nAE = Number of adverse events. Percentages are based on number of subjects in safety population in each treatment group.

Program: xxxxxx.sas

Filename

Programming Note: This table will continue for SOC and PT.

Page x of y Source:


Protocol 208821 Program Run Date: DDMMMYYYY

# Listing 16.1.7 Randomization Information All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

| Subject<br>Number | Age/Sex [1] | Randomization<br>Number | Planned Randomized<br>Treatment | Actual Treatment<br>Received | Date of Randomization |
|---|---|---|---|---|---|
| xxxxxx | xx/M | xxxx | Theraflu Powder | Theraflu Powder | DDMMMYYY |

---

[1] Age in years; Sex: M = Male

The block size of X was used for this randomization.

Page x of y
Program: xxxxxx.sas
Source: Filename

Programming Note: Block size information will be added after un-blinding of the treatment code.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.1.1 Subject Disposition All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject<br>Number | Age/Sex [1] | Screening Date | Date/Time of<br>Study Treatment<br>Administration | Date of Subject<br>Completion/<br>Withdrawal | Subject<br>Withdrawn from<br>Study? | Primary Reason for<br>Withdrawal | Further<br>Details [2] |
|---|---|---|---|---|---|---|---|
| xxxxx | xx/M | DDMMMYYYY | DDMMMYYYY/HH:MM | DDMMMYYYY | No | | |
| xxxxxx | xx/M | DDMMMYYYY | DDMMMYYYY/HH:MM | DDMMMYYYY | Yes | Protocol Violations | xxxxxx |

Page x of y
Program: xxxxxx.sas
Source: Filename

<sup>[1]</sup> Age in years; Sex: M = Male

<sup>[2]</sup> Further details of reasons for withdrawal.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.1.2 Subject Disposition Non-Randomized Subjects

Study Population: Non-Randomized Subjects (N = xx)

| Subject Number | Age/Sex [1] | Screening Date | Reason for Screen Failure | Further Details |
|---|---|---|---|---|
| XXXXXX | xx/M | DDMMMYYYY | Withdrawal Consent | XXXXXX |

[1] Age in years; Sex: M = Male.

Page x of y
Program: xxxxxx.sas
Source: Filename


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.2.1
Major Protocol Deviations
All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject Number Age/Sex [1] | | Visit(s)Excluded from<br>Scintigraphy Population | Deviation Reason |
|---|---|---|---|
| xxxxxx | xx/M | Visit 3 | Inclusion criteria |
| | | | Inclusion criteria |
| | | | XXXXXX |

[1] Age in years; Sex: M = Male.

Page x of y
Program: xxxxxx.sas Source: Filename

Programming Note: This listing is based on details in the population definition document.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.2.2 Minor Protocol Deviations All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject Number | Age/Sex<br>[1] | Visit | Deviation<br>Sequence | Date of Deviation | Deviation Type | Deviation Description |
|---|---|---|---|---|---|---|
| xxxxxx | xx/M | Visit 1 | 1 | DDMMMYYYY | xxxxxx | xxxxxx |

[1] Age in years; Sex: M = Male.

Page x of y
Program: xxxxxx.sas
Source: Filename


Protocol 208821 Program Run Date: DDMMMYYYY

# Listing 16.2.3.1 Exclusions from Analysis Population All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject Number | Age/Sex[1] | Safety Population | Scintigraphy Analysis Population |
|---|---|---|---|
| xxxxxx | xx/M | No | No |

[1] Age in years; Sex: M = Male.

Page x of y
Program: xxxxxx.sas
Source: Filename

Programming Note: This listing is based on details in the population definition document.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.4.1
Demographic Characteristics
All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject Number | Year of Birth | Age (years) | Sex | Height (cm) |
|----------------|---------------|-------------|------|-------------|
| xxxxxx | YYYY | XX | Male | XXX |

---

[1] Age in years; Sex: M = Male.

Page x of y
Program: xxxxxx.sas
Source: Filename


Protocol 208821 Program Run Date: DDMMMYYYY

#### Listing 16.2.4.2 Medical History All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject Number | Age/Sex [1] | Any Medical<br>Conditions? | Medical Condition | Start Date | Ongoing? | End Date |
|---|---|---|---|---|---|---|
| xxxxxx | xx/M | Yes | xxxxx | DDMMMYYYY | No | DDMMMYYYY |
| xxxxxx | xx/M | Yes | xxxxxx | DDMMMYYYY | Yes | |

[1] Age in years; Sex: M = Male.

Program: xxxxxx.sas

Page x of y

Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.5.1 Prior Medications All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject<br>Number | Age/Sex [1] | Drug Name<br>[GSK Drug<br>Synonym] | Reason for<br>Medication | Route of<br>Administration | Dose per<br>Administration<br>(Unit) | Frequency | Start Date<br>(Study Day<br>[2]) | End Date |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xx/M | xxxxxx<br>[xxxxxx] | xxxxx | xxxxxx | xxxxxx (xx) | xxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY |

---

<sup>[1]</sup> Age in years; Sex: M = Male.

<sup>[2]</sup> Study day is relative to the date of study treatment administration.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.5.2 Concomitant Medications All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject<br>Number | Age/Sex [1] | Drug Name<br>[GSK Drug<br>Synonym] | Reason for<br>Medication | Route of<br>Administration | Dose per<br>Administration<br>(Unit) | Frequency | Start Date<br>(Study Day<br>[2]) | Ongoing/<br>End Date |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xx/M | xxxxxx<br>[xxxxxx] | xxxxx | xxxxx | xxxxxx (xx) | xxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY |
| xxxxxx | xx/M | xxxxxx<br>[xxxxxx] | xxxxx | xxxxxx | xxxxxx (xx) | xxxxx | DDMMMYYYY<br>(xx) | Ongoing |

[1] Age in years; Sex: M = Male.

<sup>[2]</sup> Study day is relative to the date of study treatment administration.


Protocol 208821 Program Run Date: DDMMMYYYY

# Listing 16.2.6.1 Time to Onset and Completion of Gastric Emptying Scintigraphy Analysis Population

Study Population: Scintigraphy Analysis Population (N = xx)
Treatment Group: Therafly Powder

| Treatment G | roup: Theraflu Po | owder | | | | | |
|---|---|---|---|---|---|---|---|
| Subject<br>Number | Age/Sex [1] | Was<br>Scintigraphy<br>Image<br>Acquisition<br>Done? | Date<br>Scintigraphic<br>Acquisition<br>Started | Start Time of<br>Scintigraphic<br>Acquisition | End Time of<br>Scintigraphic<br>Acquisition | Gastric Emptying<br>Onset Time (min) | Gastric Emptying<br>Completion (min) |
| xxxxxx | xx/M | Yes | DDMMMYYYY | нн:мм | HH:MM | xxx | xxx |
| xxxxx | xx/M | Yes | DDMMMYYYY | HH:MM | HH:MM | xxx | XXX |

[1] Age in years; Sex: M = Male.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.7.1
All Adverse Events
All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject<br>Number | Age/Sex<br>[1] | Adverse Event<br>(Preferred Term)<br>[System Organ<br>Class] | Start Date<br>/Study<br>Day[2] | Start<br>Time | End<br>Date | End<br>Time | Frequency<br>/Intensit<br>y[3] | Related<br>to Study<br>Product? | Action<br>Taken re<br>Study<br>Product | Outcome | Serious? | Withdrew<br>?[4] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xx/M | xxxxxx<br>(xxxxxx)<br>[xxxxxx] | DDMMMYYYY/<br>xx | нн:мм | DDMMMY<br>YYY | HH:MM | INT/MILD | No | Not<br>Applicab<br>le | Recovere<br>d/Resolv<br>ed | No | No |

[1] Age in years; Sex: M = Male.

- [2] Study day is the day relative to start of treatment, day 1 being the day of first treatment.
- [3] INT = Intermittent and SGLE = Single Episode.
- [4] Did subject withdraw from study as a result of this adverse event?

Program: xxxxxx.sas

Programming Note: For Listing 16.2.7.1.2:

- Repeat the same layout for listing 16.2.7.1.2
- Population should be used 'Non randomized Subjects'
- The fourth column should be only 'Start Date (take out Study Day)'

Page x of y

Source: Filename


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.8.1.1
Laboratory Test: Urine Drug Screening
All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject Num | per Age/Sex [1] | Visit | Was Urine Sample<br>Collected at the<br>visit? | Date and Time Urine<br>Sample Collected | Result of Urine<br>Screening | Result of Urine Cotinine<br>Screening |
|---|---|---|---|---|---|---|
| ***** | xx/M | Visit 1 | Yes | DDMMMYYYY/HH:MM | Positive | Not Done: xxxxx |

---

---

[1] Age in years; Sex: M = Male.

Program: xxxxxx.sas


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.8.1.2
Laboratory Test: Breath Alcohol Screening
All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Number | | | Alcohol Screening<br>Performed? | | | (Unit) |
|---|---|---|---|---|---|---|
| xxxxxx | xx/M | Visit 1 | Yes | DDMMMYYYY/HH:MM | Positive | x.xxx (% BAC) |

---

\_\_\_

[1] Age in years; Sex: M = Male.

Program: xxxxxx.sas

Programming Note: This listing will be generated for all scheduled visits.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.8.2 Laboratory Test: Urinalysis All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject<br>Number | Age/Sex [1] | Visit | Was Urinalysis<br>Test Performed? | Date Visit | Parameters | Result |
|---|---|---|---|---|---|---|
| xxxxx | xx/M | Visit 1 | Yes | DDMMMYYYY | Specific Gravity pH Bilirubin Ketones Occult Blood Protein Nitrite Leukocyte Esterase | x.xxx<br>xx.x<br>Positive<br>Positive<br>Positive<br>Negative<br>Negative<br>Positive |

Page x of y Source: Filename

Program: xxxxxx.sas

Programming Note: This listing will be generated for all scheduled visits.

<sup>[1]</sup> Age in years; Sex: M = Male.


Protocol 208821 Program Run Date: DDMMMYYYY

> Listing 16.2.8.3 Laboratory Test: Microscopy All Randomized Subjects

Study Population: All Randomized Subjects (N = xx) Treatment Group: Theraflu Powder

| | | Examination Performed? | | | | Laboratory<br>Value |
|---|---|---|---|---|---|---|
| xx/M | Visit 1 | Yes | DDMMMYYYY | White Blood Cell | None Seen (< or = 5/HPF) | |
| | | | | Red Blood Cell | None Seen (< or = 2/HPF) | |
| | | | | Squamous Epithelial Cells | Seen | XXXXXX |
| | | | | Bacteria | Seen | XXXXXX |
| | | | | Amorphous Sediment | None Seen (/HPF) | |
| | | | | Hyaline Cast | None Seen (/LPF) | |
| | xx/M | | | | Red Blood Cell Squamous Epithelial Cells Bacteria Amorphous Sediment Hyaline Cast | = 5/HPF) Red Blood Cell None Seen (< or = 2/HPF) Squamous Epithelial Cells Bacteria Amorphous Sediment None Seen (/HPF) Hyaline Cast None Seen (/LPF) |

[1] Age in years; Sex: M = Male.

Program: xxxxxx.sas

Programming Note: This listing will be generated for all scheduled visits.


Protocol 208821 Program Run Date: DDMMMYYYY

# Listing 16.2.8.4 Laboratory Test: Serum Chemistry All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject<br>Number | Age/Sex [1] | Visit | Was Serum<br>Chemistry Test<br>Performed? | Date Visit | Parameters [Unit] | Result | High/Low<br>Categorization |
|---|---|---|---|---|---|---|---|
| xxxxxx | xx/M | Visit 1 | Yes | DDMMMYYYY | Glucose (fasting) [mg/dL] Urea Nitrogen (BUN) [mg/dL] | xxx | Low |
| | | | | | Creatinine [mg/dL] | XX<br>X.XX | High<br>Normal |
| | | | | | Sodium [mmol/L] | XXX | Normal |

---

---

Program: xxxxxx.sas

Programming Note: This listing will be generated for all scheduled visits and parameters.

<sup>[1]</sup> Age in years; Sex: M = Male.


Protocol 208821 Program Run Date: DDMMMYYYY

> Listing 16.2.8.5 Laboratory Test: Hematology All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)
Treatment Group: Theraflu Powder

| Subject<br>Number | Age/Sex [1] | Visit | Was Hematology<br>Tests Performed? | Date Visit | Parameters [Unit] | Result | High/Low<br>Categorization |
|---|---|---|---|---|---|---|---|
| xxxxxx | xx/M | Visit 1 | Yes | DDMMMYYYY | White Blood Cell (WBC) Count [Thousand/uL] | xx.x | Low |
| | | | | | Red Blood Cell (RBC) Count [Million/uL] | x.xx | High |
| | | | | | Hemoglobin [g/dL] | XX.X | Normal |
| | | | | | Hematocrit [%] | XX.X | Normal |

Program: xxxxxx.sas

Programming Note: This listing will be generated for all scheduled visits and parameters.

<sup>[1]</sup> Age in years; Sex: M = Male.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.8.6 Laboratory Test: Virology All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject<br>Number | Age/Sex [1] | Visit | Was Virology<br>Examination<br>Performed? | Date Visit | Parameters | Result |
|---|---|---|---|---|---|---|
| xxxxx | xx/M | Visit 1 | Yes | DDMMMYYYY | Hepatitis B Core AB Total<br>Hepatitis B Surface Antigen<br>Hepatitis C Antibody<br>HIV Antigen/Antibody | Non-Reactive<br>Reactive<br>Non-Reactive<br>Non-Reactive |

---

---

Program: xxxxxx.sas

<sup>[1]</sup> Age in years; Sex: M = Male.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.8.7 Listing of Normal Ranges for Laboratory Tests

| Gender | Age Group (Years) | Reference Range | |
|---|---|---|---|
| | | Low | High |
| Male | 18 | 12.0 | 16.9 |
| | 19 - 133 | 13.2 | 17.1 |
| Female | 18 | 11.5 | 15.3 |
| | 19 - 133 | 11.7 | 15.5 |
| | Male | Male 18 19 - 133 Female 18 | Male 18 12.0 13.2 Female 18 11.5 |

Program: xxxxxx.sas Page x of y


Protocol 208821 Program Run Date: DDMMMYYYY

> Listing 16.2.9.1 Vital Signs All Randomized Subjects

Study Population: All Randomized Subjects (N = xx) Treatment Group: Theraflu Powder

| Subject Number | Age/Sex [1] | Visit | Date and Time of<br>Assessment | Parameters (Unit) | Result |
|---|---|---|---|---|---|
| xxxxx | xx/M | Visit 1 | DDMMMYYYY/HH:MM | Weight (kg) | xxx.x |
| | | | | Body mass index (kg/m²) Systolic blood pressure (mmHg) Diastolic blood pressure (mmHg) Pulse rate (beats/min) Oral temperature (C) Respiratory rate (breaths/min) | xxxxx.x<br>xxx<br>xxx<br>xxx<br>xxx<br>xxx.x |

Page x of y Source: Filename

Program: xxxxxx.sas

Programming Note: This listing will be generated for all scheduled visits.

<sup>[1]</sup> Age in years; Sex: M = Male.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.9.2
Physical Examination
All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Subject Number | Age/Sex<br>[1] | Visit | Date of Visit | Parameter | Result | Details |
|---|---|---|---|---|---|---|
| xxxxxx | xx/M | Visit 1 | DDMMMYYYY | Head | Normal | |
| | | | | Ear | Abnormal | XXXXXX |
| | | | | Eyes | Abnormal, Clinically Significant | XXXXXX |
| | | | | Nose | Normal | |
| | | | | Mouth | Normal | |
| | | | | Skin | Normal | |
| | | | | Lung Examinations | Normal | |

<sup>[1]</sup> Age in years; Sex: M = Male.

Page x of y
Program: xxxxxx.sas
Source: Filename

Programming Note: This listing will be generated for all scheduled visits and parameters.


Protocol 208821 Program Run Date: DDMMMYYYY

Listing 16.2.9.3 12 Lead ECG at Screening All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| ubject Number | Age/Sex [1] | Date and Time of<br>Assessment | Parameters (Unit) | Result | Interpretation of ECG | Details |
|---|---|---|---|---|---|---|
| xxxxx | xx/M | DDMMMYYYY/HH:MM | Ventricular rate (beats/min) | XXX | Normal | |
| | | | QRS interval (msec) | XXX | | |
| | | | PR interval (msec) | XXX | | |
| | | | QT interval (msec) | XXX | | |
| | | | QTcF interval (msec) | XXX | | |

[1] Age in years; Sex: M = Male.


| D11 000001 | D D D. I DDMANUUU |
|-----------------|-----------------------------|
| Protocol 208821 | Program Run Date: DDMMMYYYY |

Listing 16.2.9.4 Weight (kg) and Body Mass Index (kg/ $m^2$ ) All Randomized Subjects

All Randomized Subjects

Study Population: All Randomized Subjects (N = xx)

Treatment Group: Theraflu Powder

| Treatment Group: | Therallu Powde | Ľ. | | | |
|---|---|---|---|---|---|
| Subject Number | r Age/Sex [1] | Visit | Date of Visit | Weight (kg) | Body Mass Index (kg/m²) |
| xxxxxx | xx/M | Visit 1 | DDMMMYYYY | XX.X | xxx.x |

---

[1] Age in years; Sex: M = Male.


Protocol 208821 Program Run Date: DDMMMYYYY

Figure 14.2.3 Plot of Mean ( $\pm$ SD) for Amount Remaining in the Stomach Over Time Scintigraphy Analysis Population

Study Population: Scintigraphy Analysis Population (N = xx)



Page x of y
Program: xxxxxx.sas
Source: Filename

Programming Note: Similar figure (Figure 14.2.4) will be generated for parameter "Sectional Areas under the Gastric Emptying Curve".